CLINICAL TRIAL: NCT06823687
Title: The Effect of Virtual Reality Glasses on Applied During Thyroid Fine Needle Aspiration Biopsy on Anxiety Level, Pain Intensity and Patient Satisfaction
Brief Title: Virtual Reality Glasses on Applied During Thyroid Fine Needle Aspiration Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, Principal Investigator, Istanbul Sabahattin Zaim University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023/06
Record Dates: First submitted 2025-02-02; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Nodule
Keywords: Thyroid Fine Needle Aspiration Biopsy
MeSH Terms: conditions — Thyroid Nodule | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality glasses (Experimental): Virtual reality glasses Beginning 1-2 minute before the start of the procedure, the patients will be watched (5-10 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses, with a music background, licensed product.
  Interventions: Other: Virtual reality glasses
- Control grups (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Virtual reality glasses — Virtual reality glasses Beginning 1-2 minute before the start of the procedure, the patients will be watched (5-10 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses, with a music background, licensed product.
  Other Names: Control group
  Arms: Virtual reality glasses

SUMMARY:
The Effect of Virtual Reality Glasses on Applied During Thyroid Fine Needle Aspiration Biopsy on Anxiety Level, Pain Intensity and Patient Satisfaction

DETAILED DESCRIPTION:
Beginning 1-2 minute before the start of the procedure, the patients will be watched (5-10 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Ability to communicate adequately
* Volunteering to participate in the research

Exclusion Criteria:

* Those with psychiatric problems
* Being unconscious

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline, pre-intervention (Before Thyroid Fine Needle Aspiration Biopsy)
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. VAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
Visual Analog Scale | Immediately after the intervention (Thyroid Fine Needle Aspiration Biopsy)
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. VAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
State-trait anxiety inventory (STAI FORM TX-1) | Baseline, pre-intervention (Before Thyroid Fine Needle Aspiration Biopsy)
  State anxiety refers to transient emotional reactions manifested by the individual to on constant situations with varying intensity depending on the situation. In situations where the individual perceives the stressful situation as a threat, the level of "state anxiety" is high and in situations where this danger is not perceived as threatening, the level of state anxiety is low. The state anxiety inventory requires the individual to describe how they feel at a given moment and under certain circumstances, taking into account their feelings about the situation in which they are in. It measures the state of the individual, that is, the level of anxiety in which they are currently in. The intensity of the instantaneous stress, anxiety, and excitement responses caused by conditions increases or decreases over time. Individuals respond to the items on the inventory based on the degree of severity of their emotions at the moment.
State-trait anxiety inventory (STAI FORM TX-1) | Immediately after the intervention (Thyroid Fine Needle Aspiration Biopsy)
  State anxiety refers to transient emotional reactions manifested by the individual to on constant situations with varying intensity depending on the situation. In situations where the individual perceives the stressful situation as a threat, the level of "state anxiety" is high and in situations where this danger is not perceived as threatening, the level of state anxiety is low. The state anxiety inventory requires the individual to describe how they feel at a given moment and under certain circumstances, taking into account their feelings about the situation in which they are in. It measures the state of the individual, that is, the level of anxiety in which they are currently in. The intensity of the instantaneous stress, anxiety, and excitement responses caused by conditions increases or decreases over time. Individuals respond to the items on the inventory based on the degree of severity of their emotions at the moment.

SECONDARY OUTCOMES:
Physiological Symptoms of Anxiety Follow-up Form | Baseline, pre-intervention (Before Thyroid Fine Needle Aspiration Biopsy)
  This form was created by the researcher to record blood pressure, heart rate, respiratory rate and peripheral oxygen saturation (SpO2) value.
Physiological Symptoms of Anxiety Follow-up Form | Immediately after the intervention (Thyroid Fine Needle Aspiration Biopsy)
  This form was created by the researcher to record blood pressure, heart rate, respiratory rate and peripheral oxygen saturation (SpO2) value.
Virtual Reality Glasses Application Satisfaction Form | Immediately after the intervention (Thyroid Fine Needle Aspiration Biopsy)
  In this form, there are questions prepared in line with the relevant literature in order to determine the satisfaction with the video watched with virtual reality glasses.

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Özer, Principal Investigator — İstanbul Sabahattin Zaim Üniversitesi
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toraman RL, Eskici Ilgin V. Effect of Virtual Reality Glasses Application on Pain, Anxiety, and Patient Satisfaction During a Transrectal Prostate Biopsy: A Randomized Controlled Trial. Biol Res Nurs. 2024 Oct;26(4):485-497. doi: 10.1177/10998004241236154. Epub 2024 Feb 28. PMID 38418943